CLINICAL TRIAL: NCT00993590
Title: Mobile CHESS Research on Emergency Medical Services for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: M-2008-1234; 5R01NR010241 (NIH)
Record Dates: First submitted 2009-10-08; First posted 2009-10-12 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
Keywords: Persistent asthma; Asthma related emergency room visits; Asthma control, adolescents; Adherence, asthma control medications
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- M CHESS group (Experimental): The intervention group will receive access for 12 months to M-CHESS via a smartphone to: (1) contact their case managers and primary provider; (2) communicate with the managed care organization case managers; (3) communicate with peers; (4) share information about changes in health status; (5) receive reminders to take medications and complete medical follow-up; (6) receive feedback on use of their asthma action plan; (7) receive tailored inquiries and insights regarding attendance or use of asthma resources; and (8) access audio and video versions of asthma educational materials and lower reading level versions of text materials; (9) provide monthly study outcome data monthly for 12 months.
  Interventions: Behavioral: M CHESS
- Control group (Active Comparator): The control group will receive standard care plus a smartphone for 12 months; they will provide study outcome data monthly for the next 12 months.
  Interventions: Behavioral: M CHESS

INTERVENTIONS:
Behavioral: M CHESS — Smartphone with access to MCHESS, an asthma control system that provides easy-to-access, just-in-time information and support.

SUMMARY:
The primary aims are to test whether an asthma care management system (M-CHESS) delivered via a smartphone (cellular phone with internet access) can support low income teenagers (ages 12-18) with significant asthma and can improve asthma control and reduce asthma-related emergency or urgent care visits and hospitalizations. Secondary aims include whether M-CHESS increases adherence to asthma control medication and reduces absenteeism from school, work or an event they wanted to attend.

DETAILED DESCRIPTION:
Four hundred Milwaukee Medicaid recipients (ages 12-18), with an asthma-related emergency care visit or hospitalization in the last twelve months, will be recruited through their managed care organization (MCO). They will be randomly assigned to one of two study arms and will participate in a 12-month intervention plus a 12-month follow-up period. Subjects in the control group will receive a smartphone with internet access & text messaging service. These devices will provide the ability to collect smartphone use data electronically. The experimental group will also receive the same smartphone devices (with internet access and text messaging service and ability to collect usedata. In addition the experimental group will have access to the Mobile CHESS (M-CHESS) interface. The M-CHESS smartphone interface features an interactive, internet based asthma education program, peer support mechanisms and automated reminders for asthma control medicines and data collection.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ranging in age from 12-18:

  * These study candidates will have had an asthma related emergency care visit or hospitalization in the last 12 months and fit the following characteristics: an ICD-9 code 493.XX and have filled one or more prescription(s) for an asthma medication (short acting beta agonist, oral corticosteroid, inhaled or nebulized corticosteroid, long-acting beta agonist, xanthine, or leukotriene modifier).
  * They also must receive medical care from one of the two participating managed care organizations involved in our study.

Exclusion Criteria:

* Other chronic pulmonary disorders such as cystic fibrosis, ABPA, or bronchopulmonary dysplasia.
* Developmental/cognitive/sensory disabilities.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 219 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Asthma control test (ACT®) scores. | One year.
Asthma-related healthcare utilization. | One year.

SECONDARY OUTCOMES:
School absenteeism. | One year.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Managed Health Services, Milwaukee, Wisconsin
  - United Healthcare, Milwaukee, Wisconsin

REFERENCES:
- See also: Related Info — http://chess.wisc.edu/chess/projects/MCHESS_EMS.aspx